CLINICAL TRIAL: NCT07351838
Title: Prognosis and Risk Stratification in Non-dilated Left Ventricular Cardiomyopathy : Cardiac MRI Insights for Better Outcomes
Brief Title: Cardiac Magnetic Resonance for Risk Stratification in Non-dilated Left Ventricular Cardiomyopathy
Status: Recruiting | Type: Observational
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Minjie Lu, Director of Magnetic Resonance Imaging, Chinese Academy of Medical Sciences, Fuwai Hospital
Other Study IDs: CMRNDLVC
Record Dates: First submitted 2025-12-29; First posted 2026-01-20 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-12

CONDITIONS: Non-ischemic Cardiomyopathy
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NDLVC
  Interventions: Other: No intervention; Observational study

INTERVENTIONS:
Other: No intervention; Observational study — No intervention; Observational study

SUMMARY:
Non-dilated left ventricular cardiomyopathy (NDLVC), a newly defined cardiomyopathy subtype characterized by non-ischemic myocardial abnormalities without left ventricular dilation, poses challenges in prognosis assessment and risk stratification. This is a retrospective observational study aiming to explore the prognostic value of cardiac magnetic resonance (CMR) findings and identify key risk factors for adverse cardiovascular outcomes in patients with NDLVC.

We will retrospectively enroll patients diagnosed with NDLVC who underwent CMR examination at the study institution during the predefined study period. CMR parameters, including left ventricular ejection fraction (LVEF), late gadolinium enhancement (LGE) patterns, myocardial strain, and the extent of myocardial fibrosis or fatty replacement, will be extracted and analyzed. The primary endpoint is a composite of major adverse cardiovascular events (MACE), including all-cause mortality, heart transplantation, or left ventricular assist device (LVAD) implantation.

The study intends to clarify the association between specific CMR features and long-term prognosis in NDLVC patients, thereby establishing a CMR-based risk stratification strategy to guide clinical decision-making and improve patient outcomes. Given the retrospective nature, data will be collected from electronic medical records and CMR databases, with ethical approval obtained prior to study initiation.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 16 years;
* indexed left ventricular end-diastolic volume (LVEDVi) <96 mL/m2 in females and <105 mL/m2 in males at baseline cardiac magnetic resonance (CMR);
* either left ventricular ejection fraction (LVEF) <50% and/or non-ischemic left ventricular (LV) scar/fatty replacement at baseline cardiac magnetic resonance.

Exclusion Criteria:

* lacked enhanced CMR images due to contraindications for receiving gadolinium contrast, such as severe renal disease;
* ischemic heart disease, defined as stenosis of >50% in a major epicardial coronary artery underwent coronary computed tomography angiography or coronary angiography, ischemic late gadolinium enhancement (LGE) pattern on CMR indicating prior infarction, or prior coronary revascularization;
* abnormal loading conditions, defined as moderate to severe valvular heart diseases, congenital heart diseases, uncontrolled hypertension;
* systemic rheumatologic diseases or sarcoidosis;
* diagnostic criteria for other cardiomyopathies according to the European Society of Cardiology (ESC) definitions.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Non-dilated left ventricular cardiomyopathy (NDLVC), formally recognized in the 2023 ESC guidelines as a distinct entity,1 encapsulates patients with non-ischemic fibrosis or fatty replacement or isolated systolic dysfunction without ventricular dilatation.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2010-01-01 (Actual); Primary Completion 2028-12-30 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
major hard cardiac event | From date of randomization until death, heart transplantation, implantation of a ventricular assist device, or the last clinical follow-up available, assessed up to 100 months.
  The primary endpoint was a composite of all-cause mortality, heart transplantation, or left ventricular assist device (LVAD) implantation. The secondary endpoint was sudden cardiac death (SCD)-related events, encompassing SCD, resuscitated cardiac arrest, ventricular fibrillation or sustained ventricular tachycardia leading to hemodynamic compromise requiring cardioversion, or appropriate implantable cardioverter-defibrillator (ICD) therapy [anti-tachycardia pacing (ATP), or shock] and heart failure (HF)-related endpoints, including HF death, heart transplant, and HF hospitalization.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese Academy of Medical Sciences and Peking Union Medical College, Fuwai Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Leo I, Dellegrottaglie S, Scatteia A, Torella D, Abete R, Aquaro GD, Baggiano A, Barison A, Bogaert J, Calo' L, Camastra G, Carigi S, Carrabba N, Casavecchia G, Censi S, Cicala G, De Cecco CN, De Lazzari M, Di Giovine G, Dobrovie M, Focardi M, Fusini L, Gaibazzi N, Gismondi A, Gravina M, Guglielmo M, Lanzillo C, Lombardi M, Lorenzoni V, Lozano-Torres J, Margonato D, Martini C, Marzo F, Masci PG, Masi A, Moro C, Muscogiuri G, Mushtaq S, Nese A, Palumbo A, Pavon AG, Pedrotti P, Perazzolo Marra M, Pradella S, Presicci C, Rabbat MG, Raineri C, Rodriguez-Palomares JF, Sbarbati S, Schoepf UJ, Squeri A, Sverzellati N, Symons R, Tat E, Timpani M, Todiere G, Valentini A, Varga-Szemes A, Volpe A, Guaricci AI, Schwitter J, Pontone G. CarDiac magnEtic Resonance for prophylactic Implantable cardioVerter defibrillAtor ThErapy in Non-Dilated Left Ventricular Cardiomyopathy: a sub-study from the DERIVATE registry. Eur Heart J Cardiovasc Imaging. 2025 Jun 30;26(7):1233-1241. doi: 10.1093/ehjci/jeaf043. PMID 39899463
- [Result] Castrichini M, De Luca A, De Angelis G, Neves R, Paldino A, Dal Ferro M, Barbati G, Medo K, Barison A, Grigoratos C, Gigli M, Stolfo D, Brun F, Groves DW, Quaife R, Eldemire R, Graw S, Addison J, Todiere G, Gueli IA, Botto N, Emdin M, Aquaro GD, Garmany R, Pereira NL, Taylor MRG, Ackerman MJ, Sinagra G, Mestroni L, Giudicessi JR, Merlo M. Magnetic Resonance Imaging Characterization and Clinical Outcomes of Dilated and Arrhythmogenic Left Ventricular Cardiomyopathies. J Am Coll Cardiol. 2024 May 14;83(19):1841-1851. doi: 10.1016/j.jacc.2024.02.041. PMID 38719365
- [Result] Arbelo E, Protonotarios A, Gimeno JR, Arbustini E, Barriales-Villa R, Basso C, Bezzina CR, Biagini E, Blom NA, de Boer RA, De Winter T, Elliott PM, Flather M, Garcia-Pavia P, Haugaa KH, Ingles J, Jurcut RO, Klaassen S, Limongelli G, Loeys B, Mogensen J, Olivotto I, Pantazis A, Sharma S, Van Tintelen JP, Ware JS, Kaski JP; ESC Scientific Document Group. 2023 ESC Guidelines for the management of cardiomyopathies. Eur Heart J. 2023 Oct 1;44(37):3503-3626. doi: 10.1093/eurheartj/ehad194. No abstract available. PMID 37622657